CLINICAL TRIAL: NCT03299140
Title: Evaluation of a Prevention Program in Children and Teenagers at High Risk for Bipolar Disorder
Brief Title: Evaluation of a Prevention Program in Children and Teenagers at High Risk for Bipolar Disorder (Bipokid)
Acronym: Bipokid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment, and investigators did not want to extend the recruitment period, so study stopped at theoretical date but number of subjects not reached
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF 9359
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2017-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Children; Family Focused Therapy; CBT
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Focused Therapy (Other): Only 1 arm
  Interventions: Behavioral: Family Focused Therapy

INTERVENTIONS:
Behavioral: Family Focused Therapy

SUMMARY:
Bipolar disorder is an early onset chronic disorder. Children of bipolar parents are at high risk of developping the same disorder and/or a psychopathology. Early intervention focused on emotion and problem solving strategies could improve their prognosis.

The main objective of this trial is to evaluate the FFT (Family Focused Therapy) efficacity. Children emotional dysregulation profile will be compared before and after this CBT intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children and teenagers from 6 to 16 years-old
* At least one biological parent with bipolar disorder
* T-score CBCL-Total ≥ 60
* Written informed consent

Exclusion Criteria:

* Active severe thymic episode
* Autism spectrum disorders
* Intellectual disability

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
CBCL-DP (Child Behavior Checklist - Dysregulation Profile) score variation | up to 12 months

REFERENCES:
- [Derived] Fongaro E, Pupier F, Picot MC, Franc N, Soler M, Olie E, Maurice V, Purper-Ouakil D, Kerbage H. Changes in emotional dysregulation profile among offspring of parents with bipolar disorder: a family-based intervention pilot study. Int J Bipolar Disord. 2025 Nov 3;13(1):31. doi: 10.1186/s40345-025-00398-3. PMID 41182531